CLINICAL TRIAL: NCT04882852
Title: Validation of the Arabic Version of the Caries Specific Measure of Quality of Life Questionnaire for Children
Brief Title: Validation of the Arabic Version of the Caries Questionnaire
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Yousry, Lecturer in pediatric dentistry and dental public health department , Cairo university, Cairo University
Other Study IDs: Validation study
Record Dates: First submitted 2021-05-03; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Dental Caries in Children
Keywords: CARIES-QC ,validity ,reliability, Arabic, dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arabic is one of the most spoken languages in the world; however, the CARIES-QC questionnaire which evaluate the effect of oral diseases and disorders on children's oral health-related quality of life has not yet been validated in Arabic speaking children. So the purpose of this study was to translate the CARIES-QC into Arabic and test the measurement properties of the Arabic version of the CARIES-QC for use in children with dental caries who speaks Arabic .

DETAILED DESCRIPTION:
Dental caries is a major public health problem. It has been estimated that 621 million children in the world have untreated dental caries . Dental caries always manifests with significant pain, affecting oral health-related quality of life (OHRQoL) and well-being. Several measures were widely used to comprehensively evaluate the effect of oral diseases and disorders on children's OHRQoL. However, most of these measures were 'generic' measures, and they may fail to detect small, clinically important changes related to specific oral diseases. Gilchrist et al recently developed the Caries Impacts and Experiences Questionnaire for Children (CARIES-QC) in order to address this issue. Preliminary findings have confirmed that Caries Impacts and Experiences Questionnaire for Children measure had good reliability, validity, and responsiveness. However, The original CARIES-QC was an English measure; so appropriate translation and cultural adaptation should be done in order to be used in other culture and language.

Arabic is one of the most spoken languages in the world; however, the CARIES-QC has not yet been validated in Arabic speaking children. So the purpose of this study was to translate the CARIES-QC into Arabic and test the measurement properties of the Arabic version of the CARIES-QC for use in children with dental caries who speaks Arabic .

ELIGIBILITY:
Inclusion Criteria:

1. Child in age from 5-16 years .
2. Child with active caries
3. Child speaks Arabic.

Exclusion Criteria:

1. Child with dental traumatic injuries .
2. Child has oral mucosal diseases.
3. Child has cleft lip and or palate .
4. Child having severe medical or mental conditions.
5. Child who cannot understand the question even with help

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children with active dental caries ranging in age from 5-16 year
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
validation of Arabic version CARIES-QC questionnaire | 1 year
  cross-cultural validity and convergent validity were performed to test validity . The confirmatory factor analysis (CFA) was used to assess the cross- cultural validity.

SECONDARY OUTCOMES:
Testing reliability of the Arabic version of CARIES-QC questionnaire | 1 year
  Two methods were used to evaluate the reliability of the scale. The internal consistency was investigated by Cronbach's alpha and inter-item correlation. To analyse the test-retest reliability, the intergroup correlation coefficient (ICC) was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Mohamed, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of dentistry, Cairo university , Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided